CLINICAL TRIAL: NCT06009081
Title: A Comparıson Of Different Interventions For Neck Paın In Relation to Internet Usage Rates
Brief Title: Interventions For Neck Pain In Relation to Internet Usage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-772.02-4942
Record Dates: First submitted 2023-08-18; First posted 2023-08-24 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Internet Addiction
Keywords: addiction; internet
MeSH Terms: conditions — Internet Addiction Disorder; Behavior, Addictive | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Physiotherapists who perform and evaluate the practice are different people.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- postural exercise (Experimental): An 8-week home exercise program consisting of neck exercises was applied for group 1. The exercise program was carried out three times a week for eight weeks.
  Interventions: Behavioral: postural exercise
- aerobic exercise (Active Comparator): An 8-week walking program was planned for Group 2 using pedometer feedback as a motivational tool.
  Interventions: Behavioral: aerobic exercise

INTERVENTIONS:
Behavioral: postural exercise — The exercises consisted of 4-way neck isometric exercises and stretching exercises for the activation of deep cervical flexors (chin tuck exercise) and combined with this exercise. This protocol consisted of protocols studied in similar studies.
  Arms: postural exercise
Behavioral: aerobic exercise — The walking program was carried out daily on a flat surface with a target of 7000 steps. This goal is based on the American College of Sports Medicine reports on the minimum recommended levels of physical activity required to achieve health benefits, which includes several design elements.
  Arms: aerobic exercise

SUMMARY:
After the rapid increase in the use of the Internet in the world, it has brought some negativities.People with internet addiction describe all the time they spend without internet as worthless and they want to be on the internet with an increasing desire.

DETAILED DESCRIPTION:
Under all this information, the exercise program and walking programs that are easily added to people's lives in the study; The effects on stress and sleep levels were investigated by reducing neck pain symptoms in people with internet addiction.

ELIGIBILITY:
Inclusion Criteria:

* 20 and 25 years old, have internet addiction
* have neck pain complaints for more than three months
* low category according to the International Physical Activity Index.

Exclusion Criteria:

* Participants who had mobility limitations and neurological problems -had spinal surgery, had a traffic accident in the last three months and were injured by whiplash injury mechanism- visual and hearing impairments,
* refused to participate in the study.

Ages: 20 Months to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2023-08-18 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
internet addiction scale | 8 weeks
  Young's internet addiction scale is a 20-question self-report scale developed by Young. There are answers to the questions as "Never", "Rarely", "Sometimes", "Often", "Very often", "Constantly". According to the survey; He was defined as "Internet addict" when he scored 80 and above
Disability Index | 8 weeks
  The Neck Disability Index is a frequently used scale to evaluate neck disability in the clinic. Pain intensity assesses perceived neck pain in personal care, lifting, reading, headaches, concentration, work, driving, sleep, and leisure activities. It was determined as "0" as the best and "50" as the worst
Physical Activity Index | 8 weeks
  The International Physical Activity Index, developed to measure the physical activity levels of individuals aged 15-65, asks questions about their physical activity in the last 7 days.It has three categories: Inactive (Category 1), Minimally Active (Category 2), Very Active (Category 3).
stress scale | 8 weeks
  Perceived stress scale, this scale is used to measure stress perceptions. In this scale, which has 14 questions in total, the answers are "Never", "Almost never", "Sometimes", "Quite often", "Very often". In this test, the lowest "0" and the highest "56" points can be obtained; high values indicate the height of the stress perceived by the person .
Sleep Quality Index | 8 weeks
  Pittsburgh Sleep Quality Index, developed by Buysse et al. in 1989, consists of 24 questions evaluating sleep status in the last 1 month. A minimum score of 21 is obtained. High scores indicate poor sleep quality
anxiety scale | 8 weeks
  The Beck anxiety scale consists of four options as "Never", "Mild", "Moderate", "Severe" considering the questionnaire responses in the last week. This scale, which has a score between 0-63 points, evaluates the symptoms of anxiety and is calculated as 63 points for the worst result. If the results are lower than 21, it indicates mild anxiety, 22-35 indicates moderate anxiety, and higher than 36 indicates severe anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- HAZAL genç, Istanbul, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang X, Yang H, Zhang K, Zhang J, Lu X, Guo H, Yuan G, Zhu Z, Du J, Shi H, Jin G, Hao J, Sun Y, Su P, Zhang Z. Effects of exercise or tai chi on Internet addiction in college students and the potential role of gut microbiota: A randomized controlled trial. J Affect Disord. 2023 Apr 14;327:404-415. doi: 10.1016/j.jad.2023.02.002. Epub 2023 Feb 6. PMID 36754096